CLINICAL TRIAL: NCT03009214
Title: A Safety, Tolerability and Pharmacokinetic Dose Escalation and Expansion, Phase I/Ib Study of AMC303 as Monotherapy in Patients With Advanced or Metastatic, Malignant Solid Tumour of Epithelial Origin
Brief Title: A Safety and Pharmacokinetic Phase I/Ib Study of AMC303 in Patients With Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: amcure GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC303-01
Record Dates: First submitted 2016-11-19; First posted 2017-01-04 (Estimated); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Malignant Solid Tumor
Keywords: solid epithelial cancer; CD44v6; c-Met; VEGFR-2; RON; receptor tyrosine kinase

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AMC303 (Experimental): cohorts will receive ascending doses of AMC303 as intravenous infusion
  Planned doses are:
  0.1 mg/kg, 0.5 mg/kg, 1.5 mg/kg, 4 mg/kg, 10 mg/kg and 20 mg/kg
  Interventions: Drug: AMC303

INTERVENTIONS:
Drug: AMC303 — AMC303 is a CD44v6 inhibitor blocking receptor tyrosine kinase (RTK) pathways
  Other Names: CD44v6 inhibitor

SUMMARY:
This is a two part Phase I/Ib, open-label, non-randomized and multi-center, dose escalation study with a 3+3 design (Part 1) and an expansion cohort at the Maximum Tolerated Dose (MTD)/Recommended Phase 2 Dose (RP2D) (Part 2). If MTD is not reached in Part 1, RP2D will be determined after completion of Part 1 considering safety and tolerability, also beyond the dose limiting toxicity (DLT) period, pharmacokinetic (PK) and pharmacodynamic (PD) results.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed and documented, advanced or metastatic, accessible malignant solid tumour of epithelial origin and for which no standard therapy exists or standard therapy has failed.
2. Presence of a measurable tumour according to RECIST 1.1. criteria
3. At least 4 weeks from the completion of any previous cytotoxic chemotherapy, 6 weeks from biological therapy (monoclonal antibodies) or cancer immunotherapy (immune checkpoint modulators) or 2 weeks from targeted therapy (receptor tyrosine kinase inhibitors) at time of administration of AMC303.
4. Male or female patients, at least 18 years of age
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 - 1
6. Life expectancy > 12 weeks.
7. Adequate haematological function defined as

   * Absolute neutrophil count (ANC) > 1,500 / µL
   * Platelets > 100,000 / µL
   * Haemoglobin > 9 g /dL.
8. Adequate renal function defined as

   * Glomerular filtration rate (GFR) ≥ 50 ml/min according to local laboratory standard or
   * Serum creatinine < 1.5 mg / dL.
9. Adequate hepatic function defined as

   * Total bilirubin < 1.5x institutional upper limit of normal (ULN)
   * AST, ALT ≤ 3x institutional ULN or < 5x institutional ULN if known hepatic metastases
   * Alkaline phosphatase < 3x institutional ULN or < 5x institutional ULN if known hepatic metastases.
10. Patient may have central nervous system (CNS) involvement if metastases have been treated and are stable at least 4 weeks after completion of radiation therapy and/or surgery. Stable disease is defined as absence of new neurological symptoms, absence of the need for steroid therapy and radiographic confirmation of stable disease. Radiographic confirmation of stable disease 4 weeks after completion of radiation therapy is not required unless indicated by neurological examination.
11. All female subjects will be considered to be of childbearing potential unless they are postmenopausal (at least 12 months consecutive amenorrhea, in the appropriate age group and without other known or suspected cause), or have been sterilized surgically. For female participants and female partners of childbearing potential, willingness and able to use two forms of highly effective contraception methods (e.g. oral contraceptive and condom, intra-uterine device and condom) while on study and for 30 days after the last study treatment. For male participants or male partners of childbearing potential, willingness and able to use two forms of highly effective contraception methods (e.g. oral contraceptive and condom, intra-uterine device and condom,) while on study and for three months after the last study treatment.
12. Provision of signed Informed Consent prior to any study related procedure being performed

Exclusion Criteria:

1. Receipt of any other investigational agent within 28 days prior to first administration of AMC303. Investigational monoclonal antibodies must not be given within 6 weeks before treatment start with AMC303.
2. Enrolment in another clinical study with an investigational drug
3. Presence of residual toxicities of CTCAE Grade > 1 after prior anti-tumour therapy within 2 weeks of first treatment with AMC303 with the exception of Grade 3 alopecia and infusion site reactions
4. Severe concurrent illness or psychiatric illness/social situation that would limit compliance with study requirements
5. Anticipation of major surgical procedures within first 4 weeks of first dose
6. Pregnancy or breast-feeding as determined by a serum pregnancy test (β-HCG) at screening prior to administration of AMC303 and willingness to father a child or to become pregnant
7. Untreated acute infectious disease
8. Patient is known to be suffering from Acquired Immune Deficiency Syndrome (AIDS) or is known to be HIV seropositive without AIDS defining disease
9. Known chronic hepatitis B or C.
10. History of allergic reactions attributed to compounds of similar chemical or biological composition to AMC303.
11. Evidence of any other medical conditions that in the opinion of the investigator may interfere with the planned treatment, affect patient compliance or place the patient at high risk from treatment-related complications
12. Previous malignant disease other than the target malignancy to be investigated within the last 5 years with the exception of basal or squamous carcinoma of the skin or cervical carcinoma in situ
13. Legal incapacity or limited legal capacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2016-12; Primary Completion 2020-07-28 (Actual); Study Completion 2021-05-07 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of AMC303 | 6 months
  Number of patients with treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
Pharmacokinetic properties of AMC303 (Cmax) | 2 days
  Determine maximum plasma concentration (Cmax)
Pharmacokinetic properties of AMC303 (AUC) | 2 days
  Determine systemic exposure (AUC) after intravenous infusion
Pharmacokinetic properties of AMC303 (t1/2) | 2 days
  Determine half-life of AMC303 after intravenous infusion
Response rate of treatment with AMC303 in patients with metastatic solid tumors | 12 months
  Determination of the complete response (CR) and partial response (PR) in patients treated with AMC303

CONTACTS AND LOCATIONS:
Overall Officials: Klaus Dembowsky, MD PhD, Study Chair — amcure GmbH
Locations (7):
- Belgium (2):
  - Jules Bordet Instiut, Brussels
  - Cliniques Universitaires Saint Luc, Brussels
- Spain (5):
  - Institut Català d'Oncologia, Hospital Duran i Reynals, L'Hospitalet de Llobregat, Barcelona
  - Vall d'Hebron Institute of Oncology (VHIO), Barcelona
  - START Madrid-CIOCC, Centro Integral Oncológico Clara Campal, Madiedo
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Instituto de Investigación Sanitaria INCLIVA, Hospital Clínico de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Matzke-Ogi A, Jannasch K, Shatirishvili M, Fuchs B, Chiblak S, Morton J, Tawk B, Lindner T, Sansom O, Alves F, Warth A, Schwager C, Mier W, Kleeff J, Ponta H, Abdollahi A, Orian-Rousseau V. Inhibition of Tumor Growth and Metastasis in Pancreatic Cancer Models by Interference With CD44v6 Signaling. Gastroenterology. 2016 Feb;150(2):513-25.e10. doi: 10.1053/j.gastro.2015.10.020. Epub 2015 Oct 24. PMID 26597578
- See also: Homepage amcure — http://www.amcure.com